CLINICAL TRIAL: NCT04788199
Title: Analytical Study of Internal Hernia Following Laparoscopic Roux-eny Gastric Bypass
Brief Title: Novel Technique in Closure of Mesenteric Defects After Laparoscopic Roux-en-Y Gastric Bypass and Its Effect on Internal Hernia: a Case-control Study
Status: Completed | Type: Observational
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmed Ghanem, Principal Investigator / As. Lecturer of General Surgery, Mansoura University
Other Study IDs: R / 17.11.105
Record Dates: First submitted 2021-03-04; First posted 2021-03-09 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Bariatric Surgery
Keywords: Bypass, Gastric; Obesity, Morbid; Glue. Internal hernia; Laparoscopy.
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-closure group: Group in which mesenteric defects were not closed after laparoscopic Roux-en-Y gastric bypass.
- Closure group: Group in which mesenteric defects were closed using cyano-acrylate glue after laparoscopic Roux-en-Y gastric bypass.
  Interventions: Other: Closure of mesenteric defects using glue

INTERVENTIONS:
Other: Closure of mesenteric defects using glue — Cyano-acrylate glue is a glue known to be used in surgery as tissue adhesive.
  Groups: Closure group

SUMMARY:
This study is to investigate the rate of internal hernia after laparoscopic Rox-en-Y gastric bypass when the defects are closed using cyano-acrylate glue.

DETAILED DESCRIPTION:
Background Internal hernia complicated by bowel obstruction is a well-recognized complication of laparoscopic Roux-en-Y gastric bypass (LRYGB). The present study aims to investigate the role of cyanoacrylate glue in the prevention of internal hernia (IH) after LRYGB and compare it with the open technique of managing mesenteric defects by leaving the mesentery intact without closure of mesenteric defects. Data from six UK hospitals have been involved in this study. Operations were done under the supervision of a single senior consultant surgeon of bariatric surgery.

Methods The prospectively collected data of 813 patients with morbid obesity who underwent LRYGB were retrospectively analyzed. Patients were subdivided into two groups: group I comprising 185 patients who had the mesenteric defects closed with cyanoacrylate glue and group II comprising 628 patients who were managed by the open technique of leaving the mesentery intact without closure of the mesenteric defects.

ELIGIBILITY:
Inclusion Criteria:

* All patients who underwent antecolic LRYGB without closure of mesenteric defects using cyanoacrylate glue or without closure of the mesenteric defects.

Exclusion Criteria:

* Open RYGB, laparoscopic converted to open RYGB, laparoscopic retro-colic RYGB, laparoscopic ante-colic RYGB with closure of the defect using sutures or RYGB done for non-bariatric purposes e.g. idiopathic gastroparesis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with morbid obesity who were qualified to receive LRYGB in the period between September 2007 and January 2020
Sampling Method: Non-Probability Sample
Enrollment: 928 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with internal hernia after Laparoscopic Roux-en-Y gastric bypass | September 2007 to January 2020

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Ghanem, Principal Investigator — Mansoura Faculty of Medicine, Imperial College Healthcare NHS Trust
Locations (1):
- St. Mary's Hospital, Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No